CLINICAL TRIAL: NCT04314193
Title: The PREDMETH Trial: Effectiveness of Methotrexate Versus Prednisone as First-line Therapy for Pulmonary Sarcoidosis - A Randomized Controlled Trial
Brief Title: Effectiveness of Methotrexate Versus Prednisone as First-line Therapy for Pulmonary Sarcoidosis
Acronym: PREDMETH
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: St. Antonius Hospital (Other); Longfonds (Unknown)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL71782.078.19
Record Dates: First submitted 2020-02-24; First posted 2020-03-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: sarcoidosis; pulmonary; prednisone; methotrexate
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Methotrexate; Prednisone

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, multi-center (17 hospitals in the Netherlands), single country, non-inferiority trial.
  Randomization 1:1 to oral prednisone (start 40 mg daily, to be tapered to 10 mg daily) or oral methotrexate (15 mg weekly to be increased to 25 mg weekly) for 24 weeks. Thereafter continuation of trial for 18 months on regular treatment (investigator decision).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methotrexate (Experimental)
  Interventions: Drug: Methotrexate
- prednisone (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Methotrexate — Oral methotrexate (15 mg weekly to be increased to 25 mg weekly) for 24 weeks.
  Arms: methotrexate
Drug: Prednisone — Oral prednisone (start 40 mg daily, to be tapered to 10 mg daily) for 24 weeks.
  Arms: prednisone

SUMMARY:
This is a prospective, randomized, non-blinded, multi-center, non-inferiority trial designed to compare effectiveness and side-effects of methotrexate versus prednisone as first-line therapy for pulmonary sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem, granulomatous disorder, most commonly affecting the lungs. Symptom burden is high, and quality of life (QoL) and social participation are negatively affected. In patients with pulmonary sarcoidosis, treatment is recommended in case of significant symptoms and/or impaired or deteriorating lung function. Evidence-based treatment recommendations are limited, outdated and largely based on expert opinion.

Prednisone is currently the first-choice therapy in pulmonary sarcoidosis and leads to short-term improvement of lung function. Unfortunately, prednisone has major side-effects and is associated with impaired QoL. Methotrexate is presently considered second-line therapy, and appears to have fewer side-effects. The investigators hypothesize that first-line treatment with methotrexate is as effective as prednisone, with fewer side-effects and better QoL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis according to the ATS/ERS/WASOG criteria, in case of absent histology a diagnosis of sarcoidosis can also be established in a multidisciplinary team meeting in a sarcoidosis expert center based on a highly suggestive clinical and radiological picture.
* Age ≥18 years.
* A pulmonary indication for treatment and parenchymal involvement on X-ray or CT-scan conducted within three months before inclusion (determined by the treating physician and conform current guidelines).
* A forced vital capacity (FVC) of ≤90% of predicted, or a diffusion capacity of the lung for carbon monoxide (DLCO) ≤70% of predicted, or ≥5% FVC absolute decline/≥10% DLCO absolute decline in the past year. For pulmonary functions tests GLI reference values are used.

Exclusion Criteria:

* Any condition or circumstance that, in the opinion of the investigator, may make a subject unlikely or unable to complete the study or comply with study procedures.
* Previous immunosuppressive treatment for sarcoidosis
* Use of systemic immunosuppressive therapy within the preceding three months for another disease than sarcoidosis
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study treatment or within 90 days after the last dose in the randomized study phase. For males; planning to pro-create during the study or within 90 days after the last dose of the randomized study phase.
* Primary systemic treatment indication being an extra pulmonary location of sarcoidosis (e.g. cardiac of neurological)
* Contra-indication for methotrexate or corticosteroids:

  * severely impaired renal function (creatinine clearance <30 ml/min)
  * impaired hepatic function (serum bilirubin-value >5 mg/dl or 85,5 micromole/l)
  * bone marrow insufficiency with severe leukopenia, thrombocytopenia, or anaemia
  * severe acute or chronic infections, such as tuberculosis, HIV, parasitic infections or other immunodeficiency syndromes
  * mouth, stomach or duodenal ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 24 weeks after inclusion
  Change in hospital-measured FVC between baseline and 24 weeks

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 4 weeks
  Change in hospital-measured FVC between baseline and 4 weeks.
Forced Vital Capacity (FVC) | 16 weeks
  Change in hospital-measured FVC between baseline and 16 weeks.
Time to major pulmonary improvement measured by FVC | 24 weeks
  Time to major pulmonary improvement measured by home-measured FVC, whereby major pulmonary improvement is defined as 80% of the maximum percent predicted FVC reached anywhere during the first 24 weeks of treatment. This will be determined on the home spirometry data.
Change in FVC | 4 weeks
  The percentage of patients with a 5 and 10% improvement or decline in FVC at 4 weeks.
Change in FVC | 16 weeks
  The percentage of patients with a 5 and 10% improvement or decline in FVC at 16 weeks.
Change in FVC | 24 weeks
  The percentage of patients with a absolute 5 and 10% improvement or decline in percent predicted FVC at 24 weeks.
Change in DLCO | 4 weeks
  The percentage of patients with a 10% or > 10% improvement or decline in DLCO at 4 weeks.
Change in DLCO | 16 weeks
  The percentage of patients with a 10% or > 10% improvement or decline in DLCO at 16 weeks.
Change in DLCO | 24 weeks
  The percentage of patients with a 10% or > 10% improvement or decline in DLCO at 24 weeks.
Changes in Angiotensin-Converting Enzyme (ACE) | 2 years
  Differences in serum levels of sACE (U/ml) in serum of sarcoidosis patients before, during and after treatment
Between group changes in sACE levels during treatment | 2 years
  Differences in serum levels of sACE (U/ml) in serum of sarcoidosis patients on prednisolone versus methotrexate
Changes in soluble interleukin-2 receptor (sIL-2R) | 2 years
  Differences in serum levels of sIL-2R (U/ml) in serum of sarcoidosis patients before, during and after treatment
Between group changes in sIL-2R levels during treatment | 2 years
  Differences in serum levels of sIL-2R (U/ml) in serum of sarcoidosis patients on prednisolone versus methotrexate
Changes in extracellular vesicles during treatment | 2 years
  Differences in absolute numbers of extracellular vesicles in serum of sarcoidosis patients before, during and after treatment
Between group changes in extracellular vesicles absolute numbers | 2 years
  Differences in absolute numbers of extracellular vesicles in serum of sarcoidosis patients on prednisolone versus methotrexate
Changes in protein expression levels in extracellular vesicles during treatment | 2 years
  Differences in protein expression in extracellular vesicles in serum of sarcoidosis patients before, during and after treatment
Between group changes in protein expression levels in extracellular vesicles | 2 years
  Differences in protein expression in extracellular vesicles in serum of sarcoidosis patients on prednisolone versus methotrexate
Changes in T lymphocyte phenotypes during Treatment | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences in phenotype of T-cells (MFI) in peripheral blood of sarcoidosis patients before, during and after treatment.
Between group changes in T lymphocyte phenotypes | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences in phenotype of T-cells (MFI) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in T lymphocyte absolute cell numbers | 2 years
  Differences in the absolute numbers of T-cells (cells/ml) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in T lymphocyte absolute cell numbers | 2 years
  Differences in the absolute numbers of T-cells (cells/ml) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in the distribution of T lymphocytes during treatment | 2 years
  Differences in the frequencies of T-cells (%) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in the distribution of T lymphocytes | 2 years
  Differences in the frequencies of T-cells (%) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in dendritic cell phenotypes during Treatment | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences in phenotype of dendritic cells (MFI) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in dendritic cell phenotypes | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences in phenotype of dendritic cells (MFI) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in dendritic cell absolute cell numbers | 2 years
  Differences in the absolute numbers of dendritic cells (cells/ml) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in dendritic cell absolute cell numbers | 2 years
  Differences in the absolute numbers of dendritic cells (cells/ml) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in the distribution of dendritic cells during treatment | 2 years
  Differences in the frequencies of dendritic cells (%) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in the distribution of dendritic cells | 2 years
  Differences in the frequencies of dendritic cells (%) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in monocyte subset phenotypes during Treatment | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences in expression of monocyte specific cell surface markers on monocytes (MFI) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in monocyte subset phenotypes | 2 years
  Flow cytometry analysis will be used to determine how the frequencies and distribution of different cell subtypes change during treatment. Different phenotypes can be identified through expression of a number of cell surface markers, expression is measured in MFI (mean fluorescence intensity).
  Differences expression of monocyte specific cell surface markers on monocytes (MFI) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in monocyte absolute cell numbers | 2 years
  Differences in the absolute numbers of monocytes (cells/ml) in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in monocyte absolute cell numbers | 2 years
  Differences in the absolute numbers of monocytes (cells/ml) in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Changes in the distribution of monocytes during treatment | 2 years
  Differences in the frequencies of monocytes in peripheral blood of sarcoidosis patients before, during and after treatment
Between group changes in the distribution of monocytes | 2 years
  Differences in the frequencies of monocytes in peripheral blood of sarcoidosis patients on prednisolone versus methotrexate
Correlation between biomarkers and clinical parameters | 2 years
  The differences in percentage of biomarkers is compared with the differences in change of FVC and DLCOc.
  Biomarkers are measured in peripheral blood and include:
  * monocytes, measured by flow cytometry (MFI)
  * Th-cells, measured by flow cytometry (MFI)
  * dendritic cells, measured by flow cytometry (MFI)
  * Proteins, measured by ELISA (ng/ml)
  * Serum biomarkers (U/l)
The King's Sarcoidosis Questionnaire (KSQ) | baseline
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The King's Sarcoidosis Questionnaire (KSQ) | baseline and 4 weeks after inclusion
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The King's Sarcoidosis Questionnaire (KSQ) | baseline and 16 weeks after inclusion
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The King's Sarcoidosis Questionnaire (KSQ) | baseline and 24 weeks after inclusion
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The King's Sarcoidosis Questionnaire (KSQ) | baseline and 1 year after inclusion
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The King's Sarcoidosis Questionnaire (KSQ) | baseline and 2 years after inclusion
  The King's Sarcoidosis Questionnaire (KSQ) assesses health status in patients with sarcoidosis. It comprises 29 items in 5 subdomains: general health status, lung, medication, skin and eyes. All scores range from 0 to 100, higher scores signifying beter health status. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline and 4 weeks after inclusion
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline and 16 weeks after inclusion
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline and 24 weeks after inclusion
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline and 1 year after inclusion
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The Chronic Respiratory Questionnaire (CRQ) | baseline and 2 years after inclusion
  The Chronic Respiratory Questionnaire (CRQ) is a 20-item self-reported validated questionnaire for HRQOL in patients with chronic respiratory disease. Scores range from 0 - 100 and higher scores signifying beter health quality.The minimal clinically important difference (MCID) is 0,5 points per item. It takes about 3-5 minutes to complete.
The global rating of change scale (GRC) | baseline
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The global rating of change scale (GRC) | baseline and 4 weeks after inclusion
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The global rating of change scale (GRC) | baseline and 16 weeks after inclusion
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The global rating of change scale (GRC) | baseline and 24 weeks after inclusion
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The global rating of change scale (GRC) | baseline and 1 year after inclusion
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The global rating of change scale (GRC) | baseline and 2 years after inclusion
  The global rating of change scale (GRC) is a measure in which patients are asked to rate if their QOL is improved or deteriorated over a certain period of time on a scale from -7 to +7. It consists of one questions and takes <1 minute to complete.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline and 4 weeks after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline and 16 weeks after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline and 24 weeks after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline and 1 year after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The EuroQol five dimensions 5-level questionnaire (EQ-5D-5L) | baseline and 2 years after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
The Medical Research Council Dyspnea scale | Baseline
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The Medical Research Council Dyspnea scale | Baseline and 4 weeks after inclusion
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The Medical Research Council Dyspnea scale | Baseline and 16 weeks after inclusion
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The Medical Research Council Dyspnea scale | Baseline and 24 weeks after inclusion
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The Medical Research Council Dyspnea scale | Baseline and 1 year after inclusion
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The Medical Research Council Dyspnea scale | Baseline and 2 years after inclusion
  The Medical Research Council Dyspnea scale consists of one question measuring dyspnea on a scale from 0-5.
The fatigue assessment scale (FAS) | Baseline
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
The fatigue assessment scale (FAS) | Baseline and 4 weeks after inclusion
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
The fatigue assessment scale (FAS) | Baseline and 16 weeks after inclusion
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
The fatigue assessment scale (FAS) | Baseline and 24 weeks after inclusion
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
The fatigue assessment scale (FAS) | Baseline and 1 year after inclusion
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
The fatigue assessment scale (FAS) | Baseline and 2 years after inclusion
  The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The MCID is 4 points or a 10% lower score.
Number of patients who discontinue/switch medication | During 24 weeks
  Every week patients register whether they missed pills (and the amount of pills wasted). Discontinuation or switch of medication is registered both by patients and researchers.
Patient Experience and Satisfaction with Medication questionnaire | baseline
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient Experience and Satisfaction with Medication questionnaire | 4 weeks
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient Experience and Satisfaction with Medication questionnaire | 16 weeks
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient Experience and Satisfaction with Medication questionnaire | 24 weeks
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient Experience and Satisfaction with Medication questionnaire | 1 year
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient Experience and Satisfaction with Medication questionnaire | 2 years
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Wijsenbeek, MD PhD, Principal Investigator — Erasmus Medical Center; Marcel Veltkamp, MD PhD, Principal Investigator — St. Antonius Hospital
Locations (17):
- Netherlands (17):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia hospital, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Medical Center Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Haaglanden Medisch Centrum, Leidschendam
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
  - VieCuri Medical Center, Venlo
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahlmann V, Janssen Bonas M, Moor CC, Grutters JC, Mostard RLM, van Rijswijk HNAJ, van der Maten J, Marges ER, Moonen LAA, Overbeek MJ, Koopman B, Loth DW, Nossent EJ, Wagenaar M, Kramer H, Wielders PLML, Bonta PI, Walen S, Bogaarts BAHA, Kerstens R, Overgaauw M, Veltkamp M, Wijsenbeek MS; PREDMETH Collaborators. First-Line Treatment of Pulmonary Sarcoidosis with Prednisone or Methotrexate. N Engl J Med. 2025 Jul 17;393(3):231-242. doi: 10.1056/NEJMoa2501443. Epub 2025 May 18. PMID 40387020
- [Derived] Kahlmann V, Janssen Bonas M, Moor CC, van Moorsel CHM, Kool M, Kraaijvanger R, Grutters JC, Overgaauw M, Veltkamp M, Wijsenbeek MS; Collaborating investigators. Design of a randomized controlled trial to evaluate effectiveness of methotrexate versus prednisone as first-line treatment for pulmonary sarcoidosis: the PREDMETH study. BMC Pulm Med. 2020 Oct 19;20(1):271. doi: 10.1186/s12890-020-01290-9. PMID 33076885